CLINICAL TRIAL: NCT05516238
Title: Systematic Use of Telepsychiatry for Outpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric Research Unit, Region Zealand, Denmark (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REG-003-2021
Record Dates: First submitted 2022-05-10; First posted 2022-08-25 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Borderline Personality Disorder; Depressive Disorder; Ptsd; Anxiety Disorders
MeSH Terms: conditions — Borderline Personality Disorder; Depressive Disorder; Stress Disorders, Post-Traumatic; Anxiety Disorders | interventions — Case Management

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video group (Experimental): Case management through video format
  Interventions: Other: Case management
- In-person (Active Comparator): Case management through in person format
  Interventions: Other: Case management

INTERVENTIONS:
Other: Case management — Case management cover therapy (psychotherapy/psychoeducation), medication adjustment, training in daily living skills (supportive), and direct consultations in crises.

SUMMARY:
Implementation and evaluation of video consultation in psychiatric outpatient treatment. The study will focus on patients' experiences regarding the use of VC. The study will also examine important aspects of the telepsychiatric consultation such as therapeutic alliance, consultation content, psychopathology and satisfaction levels compared to face-to-face consultations.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* Danish-speaking.

Exclusion Criteria:

* Exclusion criteria included a diagnosis of schizophrenia or bipolar disorder, or suffering from substance abuse.
* Additionally, Participants in the VC group were excluded if they did not have a smartphone, tablet, laptop, or personal computer with a webcam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
The demand for video consultation (VC) in clinical practice. | One year
  The demand for VC is evaluated by the percentage of included participants who chose to be in the VC group and the actual use of VC consultation sessions during the study period, including the number of missed appointments and the number of times VC sessions have been converted to telephone or in-person (IP) consultations.
Patients' therapeutic alliance, assessed by working alliance inventory- client version (WAI-C) | Two months.
  Therapeutic alliance is evaluated with the mean change scores in the WAI-C questionnaire at baseline and posttreatment. Score ranging: from 12 to 84. Higher scores indicate a higher therapeutic alliance
Patients' satisfaction, assessed by client satisfaction questionnaire 8 (CSQ-8) | Two months.
  Satisfaction is evaluated with the mean change scores in the CSQ-8 questionnaire at baseline and posttreatment. Score ranging: from 8 to 32. Higher scores indicate a higher satisfaction
Patients' Symptom level, assessed by Symptom Checklist -10 (SCL-10) | Two months.
  Symptom level is evaluated with the mean change scores in the SCL-10 questionnaire at baseline and posttreatment. Score ranging: from 0 to 100. Lower score indicates lower psychological distress
Patients' well-being, assessed by World Health Organisation- Five Well-Being Index (WHO-5) | Two months.
  Well-being level is evaluated with the mean change scores in the WHO-5 questionnaire at baseline and posttreatment. Score ranging: from 0 to 100. Higher scores indicate higher well-being
Patients' function, assessed by Sheehan Disability Scale (SDS) | Two months.
  Functional impairment is evaluated with the mean change scores in the SDS questionnaire at baseline and posttreatment. Score ranging: from 0 to 30. lower scores indicate lower functional impairment
Patient recovery, assessed by INSPIRE | Two months.
  Patient recovery is evaluated with the mean change scores in the INSPIRE questionnaire at baseline and posttreatment. Score ranging: from 0 to 100. A higher score indicates higher recovery
The implementation and integration of VC in clinical practice, as assessed by a checklist developed for the case managers (CM). | One year
  The following properties are used to evaluate the implementation and integration properties:
  1. type of technology patients use for VC sessions (Smartphone/tablet or personal computer/laptop)
  2. patients' physical location during VC session (Home or outdoor)
  3. the VC sessions confidentiality (Alone or with other persons)
  4. duration of VC session
  5. the content of the VC sessions (supportive, therapy, medication management, crisis/acute or "mix" content)
  Descriptive statistics will be applied to evaluate the implementation and integration properties.
Patients' experiences regarding the use of VC | Two months
  Semistructured interviews have been conducted to evaluate participants' experience regarding the use of VC technology in clinical practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric research unit, Region Zealand,, Slagelse, Denmark

IPD SHARING:
Plan to Share IPD: No